CLINICAL TRIAL: NCT00002274
Title: An Open Label Study Regimen of Videx (2',3'-Dideoxyinosine, ddI) in Patients With Acquired Immunodeficiency Syndrome (AIDS) Exhibiting Significant Deterioration While Taking Zidovudine (Retrovir)
Brief Title: A Study of ddI in Patients With AIDS Who Become Sicker While Taking Zidovudine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 039A; 454-999-002
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2007-10-02 (Estimated); Status verified 2007-10

CONDITIONS: HIV Infections; Leukoencephalopathy, Progressive Multifocal
Keywords: Didanosine; Drugs, Investigational; Acquired Immunodeficiency Syndrome; Zidovudine
MeSH Terms: conditions — HIV Infections; Leukoencephalopathy, Progressive Multifocal; Acquired Immunodeficiency Syndrome | interventions — Didanosine

INTERVENTIONS:
Drug: Didanosine

SUMMARY:
The objective of this open-label study regimen is to make didanosine (ddI) available to patients with AIDS who are clinically deteriorating on zidovudine (AZT) and cannot enter the Phase II ddI programs due to protocol exclusion or geographic location.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Concurrent medications for treatment of complications of AIDS are allowed.
* Aerosolized pentamidine.
* Phenytoin, but with caution.
* Note:
* Extreme caution should be exercised in the use of didanosine (ddI) in any patient receiving concurrent therapies, particularly those receiving other nucleosides (e.g., ganciclovir), drugs with toxicities similar to those observed with ddI (list included under concomitant medications section of protocol), and other drugs with significant toxicities, including many drugs used for treatment of major opportunistic infections.

Patients must be:

- Not suitable for entry into ddI phase II studies by reason of inclusion or exclusion criteria or by reason of geographic location.

Able to provide signed informed consent (parent/guardian as appropriate). Available for monthly follow-up while taking ddI. Meet required baseline laboratory values within 14 days prior to initial drug dosing.

Note:

* Extreme caution should be exercised in the use of ddI in any patient receiving concomitant therapies, particularly those receiving other nucleosides (e.g., ganciclovir), drugs with toxicities similar to those observed with ddI (list included under concomitant medications section of protocol), and other drugs with significant toxicities, including many drugs used for treatment of major opportunistic infections.

Caution should also be exercised in a patient having intractable diarrhea or patients following a low-sodium diet. Physicians caring for these patients must perform clinical and laboratory evaluations every 7-10 days for the first 2 months of ddI therapy. Should any adverse effect of any severity be detected during this period of intensive clinical and laboratory monitoring, the physician must call Bristol-Myers Squibb (1-800-662-7999). If the patient continues ddI therapy, Bristol-Myers Squibb will require submission of follow-up and adverse experience report forms every 10 days. Although data are not available to fully assess the risks associated with the use of ddI in high-risk patients (for example, patients with preexisting disorders of body systems known to be adversely affected by ddI, particularly those with history of peripheral neuropathy, pancreatitis, seizure disorder, cardiac abnormalities, gout, and significant elevations of liver function test results), all such patients must have clinical and laboratory evaluations performed every 10 days and results submitted to Bristol-Myers Squibb on the case report forms provided.

Exclusion Criteria

Co-existing Condition:

Patients with any one of the following criteria are excluded:

* Received therapy in the preceding 15 days with any other antiretroviral except zidovudine (AZT).
* Taking AZT concomitantly.
* Acute pancreatitis.
* Poorly controlled seizure disorder.
* Taking phenytoin concomitantly.
* Grade B or greater peripheral neuropathy.

Concurrent Medication:

Excluded:

* Zidovudine (AZT).

Patients with any one of the following criteria are excluded:

* Received therapy in the preceding 15 days with any other antiretroviral except zidovudine (AZT).
* Taking AZT concomitantly.
* Taking phenytoin concomitantly.
* Acute pancreatitis.
* Poorly controlled seizure disorder.
* Grade B or greater peripheral neuropathy.

Prior Medication:

Excluded within 15 days of study entry:

* Any antiretroviral except zidovudine (AZT).

Required:

* Zidovudine (AZT).

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Bristol - Myers Squibb Co, Princeton, New Jersey, United States

REFERENCES:
- [Background] Abrams DI. Treatment options in zidovudine intolerance or failure. AIDS. 1994 Sep;8 Suppl 3:S3-7. doi: 10.1097/00002030-199409001-00002. PMID 7840914